CLINICAL TRIAL: NCT04092868
Title: Heparin Antagonization by Protamine in Cardiac Surgery: Pharmacokinetic/Pharmacodynamic Study
Acronym: PICS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19CH046; 2019-000859-14 (EudraCT Number)
Record Dates: First submitted 2019-09-09; First posted 2019-09-17 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Surgery Requiring Extracorporeal Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery with extracorporeal circulation: during the operation
  Intervention Blood sample :
  - Choay Heparin (pharmacokinetic) concentration: t = 5, 15, 30 minutes after the start of the heparin injection + t = 5, 30, 60 minutes after the start of extracorporeal circulation
  * protamine dosage: t = 2, 5, 8, 10 and 15 min after protamine injection
  * anti-X activity t = 0 before administration and at time 2, 5, 8, 10 and 15 min then at time 1, 3, 5, 6 and 7 hours after protamine injection
  * thrombin generation test (TGT) activity (thrombinography) : t = 2, 5, 8, 10 and 15 min after protamine injection
  Interventions: Other: Blood samples PK/ PD protamine

INTERVENTIONS:
Other: Blood samples PK/ PD protamine — PK/ PD protamine

SUMMARY:
Protamine is currently used during cardiac surgery to neutralize unfractionated heparin (UFH) at the end of extra-corporeal circulation (ECC). The optimal dose of protamine is currently unknown, and the administration of protamine is done empirically.

Protamine and UFH pharmacokinetics are characterized by a large inter-individual variability. A dose of protamine proportional to the amount of UFH administrated during the surgery may be therefore not adapted to most of the patients and exposed them to a risk of under or over dosage.

In this study, research investigators hypothesize that an accurate characterization of the pharmacokinetic/pharmacodynamic (PK/PD) relationship of protamine may help to optimize propose an optimal dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients benefiting from scheduled or emergency at the Saint-Etienne University Hospital (coronary artery bypass grafting, valve replacements, aortic dissections).

Exclusion Criteria:

* Patients with a contraindication to UFH
* Patients with a contraindication to protamine
* Patients requiring early resurgery.
* Patients receiving an injection of antithrombin III.
* Pregnant women.
* Patient for whom aprotinin use is planned during surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cardiac surgery under CEC
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
PK/PD Protamine | 1 day
  Pharmacokinetics (PK) : plasma concentration of protamine measured by liquid chromatography coupled with mass spectrometry.
  Pharmacodynamics (PD) :The effect of protamine corresponds to the kinetics of the disappearance of UFH in the blood. To do this, the investigators measure its concentration using an anti-Xa activity measurement technique.

SECONDARY OUTCOMES:
PK/PD Protamine | 1 day
  PK: evolution of protamine concentrations over time (plasma concentration of protamine measured by liquid chromatography coupled with mass spectrometry).
  PD: ts neutralizing effect evaluated by thrombinography .
postoperative blood loss: | 1 day
  quantities of blood loss in pleural and mediastinal drains during the first 24 hours postoperatively.
ratios between the amount of UFH present at the protamine injection and the dose of protamine administered. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Julien LANOISELÉE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanoiselee J, Gibert A, Gouin-Thibault I, Mansour A, Pontis A, Morizot C, Goset M, Molliex S, Morel J, Noyel P, Azarnoush K, Petrosyan A, Delavenne X, Zufferey PJ, Ollier E. Optimising protamine dosing for heparin reversal after cardiopulmonary bypass: a population pharmacokinetic-pharmacodynamic study. Br J Anaesth. 2026 Feb 3:S0007-0912(25)00892-X. doi: 10.1016/j.bja.2025.11.057. Online ahead of print. PMID 41638976